CLINICAL TRIAL: NCT05418868
Title: A Phase I, Multi-centre, Open-label, Single Dose Escalation Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Long-acting Cabotegravir Co-administered With Recombinant Human Hyaluronidase PH20 (rHuPH20) in Healthy Adult Volunteers
Brief Title: A Study to Investigate Pharmacokinetics, Safety and Tolerability of Long-Acting Cabotegravir Plus Recombinant Human Hyaluronidase PH20 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry); Janssen Sciences Ireland Unlimited Company (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 218012
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: Cabotegravir (CAB); Rilpivirine (RPV); Long-Acting Injection; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: Participants receiving CAB 200 mg/mL with rHuPH20 (Experimental): Part A of the study (CAB 200 mg/mL with rHuPh20) has been closed to further enrolment based on preliminary results.
  Interventions: Drug: Cabotegravir 200 mg/mL; Drug: rHuPH20
- Part C: Participants receiving CAB >=400 mg/mL or CAB Formulation I or CAB Formulation J (Experimental)
  Interventions: Drug: Cabotegravir >=400 mg/mL; Drug: Cabotegravir Formulation I; Drug: CAB Formulation J
- Part E: Participants receiving RPV (Experimental)
  Interventions: Drug: RPV

INTERVENTIONS:
Drug: Cabotegravir 200 mg/mL — CAB 200 mg/mL will be administered.
  Arms: Part A: Participants receiving CAB 200 mg/mL with rHuPH20
Drug: Cabotegravir >=400 mg/mL — CAB >=400 mg/mL will be administered by IM or SC injection.
  Arms: Part C: Participants receiving CAB >=400 mg/mL or CAB Formulation I or CAB Formulation J
Drug: Cabotegravir Formulation I — CAB Formulation I will be administered by IM injection.
  Arms: Part C: Participants receiving CAB >=400 mg/mL or CAB Formulation I or CAB Formulation J
Drug: CAB Formulation J — CAB Formulation J will be administered by IM injection.
  Arms: Part C: Participants receiving CAB >=400 mg/mL or CAB Formulation I or CAB Formulation J
Drug: rHuPH20 — rHuPH20 will be administered.
  Arms: Part A: Participants receiving CAB 200 mg/mL with rHuPH20
Drug: RPV — RPV will be administered by IM injection.
  Arms: Part E: Participants receiving RPV

SUMMARY:
This is an open-label, dose-escalation study to investigate the safety, tolerability and pharmacokinetics (PK) of single subcutaneous (SC) administration of long acting (LA) Cabotegravir (CAB) 200 milligrams per milliliter (mg/mL) with Recombinant Human Hyaluronidase PH20 (rHuPH20) (Part A), a single-dose or repeat-dose SC or intramuscular (IM) administration of LA CAB (greater than or equal to) >=400 mg/mL (Part C), single-dose IM administration of LA CAB Formulation I (Part C Cohort C8) and LA CAB Formulation J (Part C Cohort C11), and a single-dose or repeat-dose IM administration of rilpivirine (RPV) (Part E). Part A of the study (CAB 200 mg/mL with rHuPh20) has been closed to further enrolment based on preliminary results. Part D of the study (CAB >=400 mg/mL with rHuPH20) will not be conducted due to changes in the study design.

ELIGIBILITY:
Inclusion Criteria:

* At the time of obtaining informed consent, participants age should be greater than or equal to (>=)18 years and less than or equal to (<=) 55 years.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight >=40 kilogram (kg) and body mass index (BMI) within the range >=18 to <=32 kilogram per meter square (kg/m^2).
* Participants who are negative on a single test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (approved molecular polymerase chain reaction [PCR] laboratory or point of care test), performed on the day of admission. A negative result is required prior to the administration of study intervention on Day 1.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving written informed consent.

Exclusion Criteria:

* Current presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including participants who have required treatment for seizures within this time period.
* Positive SARS-CoV-2 polymerase chain reaction test, having signs and symptoms which in the opinion of the investigator are suggestive of coronavirus disease 2019 (COVID-19) (i.e., fever, cough etc) within 14 days of inpatient admission, or having contact with known COVID-19 positive person/s in the 14 days prior to inpatient admission.
* Human immunodeficiency virus (HIV-1 or HIV-2) infection as indicated by positive antibody/antigen test.
* History of or on-going high-risk behaviors that, in the opinion of the investigator, may put the participant at increased risk for HIV infection including, but not limited to, participants in HIV discordant relationships, or men who report current or prior unprotected anal sex with other men and those reporting prior or current injecting drug use.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Abnormal blood pressure.
* Evidence of previous myocardial infarction.
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [2nd degree or higher], Wolff- Parkinson-White [WPW] syndrome).
* Any significant arrhythmia which, in the opinion of the investigator or the medical monitor, will interfere with the safety for the individual participant.
* One or more exclusionary values for a screening Electrocardiogram (ECG).
* Alanine transaminase (ALT) >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Estimated Glomerular Filtration Rate (eGFR) <60 milliliter per minute (mL/min) using the Chronic Kidney Disease
* Improved Prediction Equations (CKD-EPI) Creatinine Equation (2021).
* Hemoglobin <12.5 gram per deciliter (g/dL) for men and <11 g/dL for women.
* Positive pre-study drug/alcohol screen.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to screening; or urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g., nicotine patches or vaporizing devices).
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for males or >7 units for females.
* Regular use of known drugs of abuse.
* Concurrent participation in another clinical trial (except imaging trials); or has participated in a clinical trial and received an investigational product within the following time period prior to the first dosing day in this study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than four (4) new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study interventions (or components thereof), a history of drug allergy or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation, including a known hypersensitivity to hyaluronidases.
* Current or anticipated need for chronic anti-coagulation therapy.
* Hereditary coagulation and platelet disorders (e.g., hemophilia or Von Willebrand disease [VWD]).
* Participant has a tattoo overlying the location of injection or an underlying skin disease or condition (e.g., infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) that, in the opinion of the investigator, may interfere with interpretation of injection site reactions or administration of study intervention.
* Any other clinical condition, behavior or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study; unable to comply with dosing requirements; or unable to comply with study visits.
* Participant who in the investigator's judgment poses a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Time of maximum observed plasma concentration (tmax) of Cabotegravir CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Area under the concentration - time curve from time zero to infinity (AUC[0-inf]) of CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Area under the concentration - time curve from time zero to time of last quantifiable concentration or 4 weeks following the injection whichever is earlier (AUC[0-t]) of CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Cohorts Part A, C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohort C10 [Part C])
Area under the concentration - time curve from time zero to last quantifiable time point or 8 weeks following the injection whichever is earlier [AUC(0-t)] | Up to end of study (Week 72 for Cohort C10 [Part C])
Plasma Concentration of CAB and RPV at Week 4 | Week 4
Plasma Concentration of CAB and RPV at Week 8 | Week 8
Plasma Concentration of CAB and RPV at Week 12 | Week 12
Plasma Concentration of CAB and RPV at Week 16 | Week 16
Plasma Concentration of CAB and RPV at Week 24 | Week 24
Plasma Concentration of RPV at Week 32 | Week 32
Plasma Concentration of CAB at Week 36 | Week 36
Plasma Concentration of RPV at Week 40 | Week 40
Plasma Concentration of CAB and RPV at Week 48 | Week 48
Plasma Concentration of CAB | At weeks 56, 64 and 72 for Cohorts C11 and C10 [Part C]
Plasma Concentration of RPV at Week 56 | Week 56
Plasma Concentration of RPV at Week 64 | Week 64
Plasma Concentration of RPV at Week 72 | Week 72
Apparent terminal phase half-life (t1/2) of CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Apparent long-acting absorption rate constant (KA-LA) of CAB and RPV | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Number of Participants with Non-serious Adverse Events (non-SAEs) and Serious Adverse Events (SAEs) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Number of Participants with AEs by Severity | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute value of Hematology parameter: Platelet count (cells per microliter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Hematology parameters: Reticulocytes (Percentage of reticulocytes) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Hematology parameters: Hematocrit (Proportion of red blood cells in blood) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Hematology parameters: Hemoglobin (Hgb) (grams per deciliter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C] , and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute value of Hematology parameter: Red Blood Cell Count (RBC) (million cells per microliter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C] , and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute value of Hematology parameter: Mean Corpuscle Volume (MCV) (Femtoliters) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C] , and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute value of Hematology parameter: Mean Corpuscle Hemoglobin (MCH) (Picograms) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Hematology parameters: Differential count of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per liter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Clinical Chemistry parameters: Glucose (fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per deciliter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Absolute values of Clinical Chemistry parameters: AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per liter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
  Clinical chemistry parameters such as Aspartate Aminotransferase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase and (SGPT), Alkaline phosphatase (ALP) and Creatinine Phosphokinase (CPK) will be analyzed.
Absolute values of Clinical chemistry parameters: Albumin and Total Protein (Grams per deciliter) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameter: Platelet count (cells per microliter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameters: Reticulocytes (Percentage of reticulocytes) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameters: Hematocrit (Proportion of red blood cells in blood) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameters: Hgb (grams per deciliter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameter: RBC Count (million cells per microliter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameter: MCV (Femtoliters) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameter: MCH (picograms) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Hematology parameters: Differential count of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (Giga cells per liter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Clinical Chemistry parameters: Glucose (fasting), BUN, Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per deciliter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Clinical Chemistry parameters: AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per liter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Change from Baseline in Clinical chemistry parameters: Albumin and Total Protein (Grams per deciliter) | Baseline (Day 1) and up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Number of participants with maximum toxicity grades increase from Baseline in hematology and clinical chemistry | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])

SECONDARY OUTCOMES:
Dose proportionality of CAB and RPV based on AUC(0-inf) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Dose proportionality of CAB and RPV based on AUC(0-t) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Dose proportionality of CAB and RPV based on Cmax | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Dose proportionality of CAB and RPV based on plasma concentration | Weeks 4, 8, 12 and 24
Number of participants with maximum post-baseline QTc values compared to baseline by category (to <=450 milliseconds (msec) or no change, to >450 msec to <=480 msec, to >480 msec to <=500 msec, and to >500 msec) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Number of participants with maximum post-baseline increase in QTc values compared to baseline based on category (increase <=30 msec, increase of 31-60 msec, and increase of >60 msec) | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline for diastolic blood pressure (DBP), systolic blood pressure (SBP) and pulse rate | Up to end of study (Week 78 for Cohorts C1 and C3 [Part C], Week 52 for Part A, Cohorts C2, C4, C5, C6, C7, C8, C9 [Part C], and Week 72 for Part E and Cohorts C10 and C11 [Part C])
  Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline will be categorized into change to low, change to within range or no change, and change to high.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (3):
- United States (3):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/